CLINICAL TRIAL: NCT03605966
Title: Developing a Method to Objectively Measure Opioid Analgesia: A Pilot Study
Brief Title: Developing a Method to Objectively Measure Opioid Analgesia
Status: Active, not recruiting | Type: Observational
Sponsor: Julia Finkel (Other)
Responsible Party: Sponsor-Investigator, Julia Finkel, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 6825
Record Dates: First submitted 2018-07-10; First posted 2018-07-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Analgesics, Antipyretics and Anti-Inflammatory Drugs Causing Adverse Effects in Therapeutic Use
Keywords: analgesia; pain; nociception; pupillometry; analgesic; opioid
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Inappropriate prescribing is the fundamental upstream driver of the opioid epidemic. Objective measures to determine the appropriateness of an opioid intervention, provide monitoring of the therapy for adequacy of dose and detection of tolerance or hyperalgesia would eliminate the subjective nature of opioid mediated pain management and obviate iatrogenic facilitation of opioid abuse. The present study is designed to objectively determine whether our device can pain type and determine analgesic efficacy thereby optimizing treatment selection and opioid management.

DETAILED DESCRIPTION:
It is generally recognized that pain assessment and management in newborns and children is an unmet need. The Center for Disease Control found that in 2012, healthcare providers wrote 259 million prescriptions for opioid painkillers contributing to an epidemic of over prescription. At the same time, medical professionals still see large amounts of pain left untreated, particularly in pediatric populations. Children are often given minimal or no analgesia for procedures that are treated much more aggressively in adults. This issue stems from the lack of an effective method of assessing and monitoring patient analgesia. Recently attempts have been made to objectively quantify pain but as of now, no effective standard exists. This pilot study utilizes pupillary reflexes to characterize opioid analgesia in pediatrics with the purpose of synthesizing the data into algorithms that detect specific conditions and provide decision support.

Pupillometry is a useful, non-invasive clinical and research tool that can provide valuable insights into the autonomic nervous system. Pupillary tests provide a convenient and simple method for evaluation of autonomic function4. In normal pupillary responsiveness, pupils should be equal in size, approximately 3-4mm in size under average light conditions, and reactive to light at >1mm of movement. The sympathetic nervous system is activated during periods of pain and stress and creates relaxation of the ciliary muscles resulting in pupillary dilation, or mydriasis. In accommodation, the parasympathetic axons that innervate the iris muscle produce constriction, or miosis. This reflex is known as the pupillary reflex dilation (PRD) and has been shown in previous studies to occur in both awake and anesthetized participants following a noxious stimulus5. This protocol will utilize these known reactions to track the response to specific neurostimulation in participants receiving opioids to determine the effect and effectiveness of the treatment.

All mu opioid agonists cause miosis (constriction of the pupil) thus reducing the constriction amplitude and constriction velocity of the pupillary light reflex (PLR). This is the one opioid side effect to which tolerance does not occur. However, the pharmacologic impact is not consistent and will vary with different drugs in the class and duration of exposure. For example, morphine and Dilaudid (hydromorphone) each produce a neuro-excitatory metabolite that causes mydriasis or dilation of the pupil and also antagonizes the parent drug, producing the clinical appearance of tolerance, requiring more drug to achieve the same effect. With other drugs of this class such as fentanyl, which is commonly administered in ICUs, mydriasis may occur due to a phenomenon called opioid induced hyperalgesia (OIH) where there is an increased sensitivity to pain, often leading to an increased dose of drug. Increasing the dosing in this situation can potentially exacerbate the issue, having a method to monitor for OIH would provide decision support to physicians and allow them to recognize and properly reconcile this issue. Evaluation of PRD in response to a 5 Hz neuro-stimulus can differentiate between these drug-related issues and disease progression. This works because opioid receptors populate the C fibers, which are stimulated with a 5 Hz frequency6,7, allowing the investigators to determine dose response relationships as well as the optimized analgesic dose and precisely determine dosing with opioid rotation. This occurs empirically during standard of care based on a trial and error approach that risks under or overdosing patients and having tolerance, dependence and OIH occur.

This pilot study is part of an ongoing effort to develop a method to objectively assess pain and its response to specific interventions. It specifically aims to develop profiles of the impact of a variety of opioids under a variety of conditions in a diverse patient population. It will allow researchers to understand better the specific impact of drugs in this class on the PLR and PRD. Data collected herein will help will evaluate the feasibility of using this approach to detect and monitor opioid analgesia and open new avenues for future research in this area.

1. Pain assessment and baseline testing
2. Standardized care where patient receives opioid dose per clinical team.
3. Testing pupillary reflexes at regular intervals and repeated pain assessments

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 7 to 21 years of age
2. The subject is receiving an opioid via bolus or a patient controlled analgesia (PCA) apparatus as part of treatment or fentanyl infusion in the pediatric intensive care unit (PICU) (generally postoperative patients).
3. The subject is willing and able to provide written informed assent/parental consent to study participation

Exclusion Criteria:

1. Eye pathology precluding pupillometry
2. For patients in the PICU, patients who are hemodynamically unstable

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who are receiving opioid as part of their standard care will be recruited from the Inpatient Pain at Children's National Medical Center (CNMC).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Pupillary Dilation Reflex AUC | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  The primary measurable outcomes for this study are the changes in the PRD area under the curve (AUC) that occur as a response to an opioid exposure. The differences are calculated by comparing the parameters from before the opioid dose to various time points after the opioid dose.

SECONDARY OUTCOMES:
Pain Assessment by Visual Analog Scale (VAS) | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  Collection of the standard Visual Analog Scale (VAS) with scores of of 1-10. A score of 10 signifies maximal pain and a score of 1 signifies no pain.
Pupillary Dilation Reflex Amplitude | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  A secondary measurable outcome for this study are the changes in the PRD amplitude that occur as a response to an opioid exposure. The differences are calculated by comparing the parameters from before the opioid dose to various time points after the opioid dose.
Changes in Pupillary Light Reflex Amplitude | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  A secondary measurable outcome for this study are the changes in the PLR amplitude that occur as a response to an opioid exposure. The differences are calculated by comparing the parameters from before the opioid dose to various time points after the opioid dose.
Changes in Pupillary Light Reflex Latency | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  A secondary measurable outcome for this study are the changes in the PLR latency that occur as a response to an opioid exposure. The differences are calculated by comparing the parameters from before the opioid dose to various time points after the opioid dose.
Changes in Pupillary Light Reflex Constriction Velocity | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  A secondary measurable outcome for this study are the changes in the PLR constriction velocity that occur as a response to an opioid exposure. The differences are calculated by comparing the parameters from before the opioid dose to various time points after the opioid dose.

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Finkel, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT03605966/Prot_SAP_000.pdf